CLINICAL TRIAL: NCT05627128
Title: Anti-Inflammatory Diet (Dieta Antiinflamatoria or DAIN in Spanish): a Crohn's Disease Management Strategy Tailored for Puerto Ricans
Brief Title: A Culturally Tailored Dietary Intervention to Treat Crohn's Disease
Acronym: DAIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Puerto Rico (Other); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Principal Investigator, Ana Maldonado-Contreras, Assitant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1250122; R-2102-05006 (Other Grant/Funding Number: The Leona M. and Harry B. Helmsley Charitable Trust)
Record Dates: First submitted 2022-10-11; First posted 2022-11-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-03

CONDITIONS: Crohn Disease
Keywords: diet; inflammation; microbiome
MeSH Terms: conditions — Crohn Disease; Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized intervention trial in adults with Crohn's disease.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All staff collecting data (e.g., dietary assessment) or assaying samples (e.g., fecal calprotectin, cytokines, sequencing) including the PI's, will be blinded to diet group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm1: Crohn's disease patients + DAIN (Experimental): Participants will have 10 weeks of DAIN intervention (From week 1 to week 10)
  Interventions: Other: DAIN
- Arm 2: Crohn's disease patients no intervention (No Intervention): Participants will continue consuming their usual diet, with no intervention

INTERVENTIONS:
Other: DAIN — Participants in the experimental arm will have access to the newly created DAIN curriculum including menus, recipes, and recorded 'how to' recipes. Participants in the experimental arm will also have once-per-week dietary counseling with DAIN-trained nutritionists and monthly cooking classes with a DAIN-trained chef.
  Arms: Arm1: Crohn's disease patients + DAIN

SUMMARY:
The goal of the study is to test the efficacy of a dietary intervention in inducing clinical response and remission for patients with Crohn's disease in a randomized controlled trial. The intervention diet: DAIN has been adapted from the Inflammatory Bowel Disease Anti-Inflammatory Diet or IBD-AID™ taking into account the food availability and preferences of Puerto Ricans. DAIN also includes traditional foods commonly consumed in the typical Puerto Rican diet while maintaining the fundamental components of the IBD-AID™.

DETAILED DESCRIPTION:
Crohn's disease is a chronic recurrent inflammatory disorder of the gastrointestinal that results from an inappropriate inflammatory response to an altered gut microbiome (i.e., dysbiosis). Diet is the main driver of microbiome composition. Diet also has been increasingly recognized as a cost-effective strategy to induce remission in pediatric and adult patients with Crohn's disease but diets that can substitute traditional and locally available foods among Puerto Ricans have not been explored. DAIN, a newly created dietary program, incorporates an extensive patient curriculum of recipes and menus adapted to the local availability and food preferences of Puerto Rican patients with Crohn's disease. This study aims to address three questions: whether DAIN a diet adapted to Puerto Rican patients with Crohn's disease, can: 1) induce clinical response and remission; 2) change the inflammatory tone, and 3) revert dysbiosis in Crohn's disease patients.

Participants will be randomized 1:1 ratio into two arms:

* Arm 1 Crohn's disease patients + DAIN (Experimental): this group of patients will participate in ten weeks of DAIN intervention (From week 1 to week 10)
* Arm 2 Crohn's disease patients no intervention (Control): this group of patients will not participate in the DAIN dietary intervention and will continue the usual diet.

Participation in the study lasts for 15 weeks with four-time points: week 0 (baseline), week 6, week 10, and week 14. At each time point, all subjects will complete a series of questionnaires to assess overall health, Crohn's disease activity, and dietary compliance. Blood and stool samples will be also collected at home at each time point. Samples will be either shipped or brought to the Research Unit at the Inflammatory Bowel Disease Clinic at the University of Puerto Rico.

The primary outcome is Improvement of health-related quality of life. Secondary outcomes are: (i) reduction of inflammation, (ii) changes in the gut microbiome, (iii) clinical response and remission,and (iii) dietary compliance.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 65 years old
* Confirmed CD diagnosis with sCDAI <450 (includes values ranging from remission, mild to moderate activity)
* Moderate to severe impaired QoL (sIBDQ<60)
* Stable doses of medications are screened; thiopurines, natalizumab, methotrexate (12 weeks), anti-tumor necrosis factor (TNF), ustekinumab, vedolizumab (8 weeks), 5-aminosalicylic acid (5-ASA) (2 weeks), steroids (1 week)
* Willingness and capacity to significantly change diet (arm 1)
* Willing and able to comply with specimen collection and other study procedures, and to complete the study

Exclusion Criteria:

* Ostomy
* Use of Specific Carbohydrate Diet of IBD-AID™ within 4 weeks of screening
* Use of prescribed probiotics within 4 weeks of screening
* > 20mg prednisone or equivalent
* Recent C. difficile colitis
* Pregnancy
* Presence of symptomatic or significant structure or history of obstruction in the past 6 months

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of health-related quality of life | Week 0, 6, 10, 14
  Improvement of health-related quality of life (increase of the short Inflammatory Bowel Disease Questionnaire score (SIBDQ)). The SIBDQ scores range between 10 and 70 points. A slightly impaired quality of life is indicated by scores from 60 to 70 points, moderately impaired quality of life from 45 to 60 points, and severely impaired quality of life from 10 to 45 points.

SECONDARY OUTCOMES:
Change of Inflammation | Week 0, 6, 10, 14
  Changes in inflammation will be determined by levels of calprotectin in stools and C-reactive protein (CRP) in the blood. Both stool and blood will be collected at each time point. Decreased levels of fecal calprotectin and CRP indicate a decrease in inflammation and vice versa.
Gut Microbiome changes | Week 0, 6, 10, 14
  Gut microbiome changes related to the dietary intervention will be assessed by metagenomic shotgun sequencing of stool samples collected at each time point.
Dietary compliance | Week 0, 6, 10, 14
  DAIN Dietary compliance will be evaluated by calculating the Healthy Eating Index (HEI) score from the assessment tools: 24-Hour Dietary Recalls (24HDRs) and Food Frequency Questionnaires, surveyed at each time point. The HEI is composed of 13 diet components: total fruits, whole fruits, total vegetables, greens and beans, dairy, total protein foods, seafood and plant proteins, fatty acids, refined grains, whole grains, sodium, added sugars, and saturated fats. A minimum number of servings per component have been established, and the scoring of the HEI components is based on these established values. The total maximum score is equal to 100. Higher values represent closer compliance with DAIN.
Clinical response and remission | Week 0, 6, 10, 14
  Clinical response and clinical remission will be assessed by reduction of the Short Crohn's Disease Activity Index or SCDAI. Scores range from 0 to 600 with different. A score less than 150 indicates remission, a score between 150-219 indicates mild activity, a score from 220 and 450 indicates moderate activity, and a score greater than 450 indicates severe activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ana L Maldonado-Contreras, PhD, Principal Investigator — University of Massachusetts Chan Medical School
Locations (2):
- University of Massachusetts Chan MedicaL School, Worcester, Massachusetts, United States
- University of Puerto Rico, San Juan, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
All sequence data generated in this trial are understood to represent community resources and will be submitted to the appropriate public database. Specifically, data will be submitted to the NCBI (https://www.ncbi.nlm.nih.gov/), lncrnadb (http://www.lncrnadb.org/), and NONCODE (http://www.noncode.org/) databases as soon as sequencing data becomes available but not later than 2 years.
  Sequence data will also include information on quality values for each sequence as well as required fields for metagenomic data. The study will be in compliance with the NIH Genomic Data Sharing (GDS).
  Materials generated under the project will be disseminated in accordance with University/ Participating institutional and NIH policies.
Time Frame: 2 years
Access Criteria: Access to databases and associated software tools generated under the project will be available for educational, research and non-profit purposes. A portal will be created on the study website whereby anyone interested in collaborating or accessing to the data may submit a request form. Publication of data shall occur during the project, if appropriate, or at the end of the project, consistent with normal scientific practices. Research data, which documents, supports and validates research findings will be made available after the main findings from the final research data set have been accepted for publication. Such research data will be redacted to prevent the disclosure of personal identifiers.